CLINICAL TRIAL: NCT02078947
Title: Optimizing Exercise Training in Prevention and Treatment of Diastolic Heart Failure- Clinical Study
Brief Title: Optimizing Exercise Training in Prevention and Treatment of Diastolic Heart Failure
Acronym: OptimEx-Clin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: European Commission (Other); University of Leipzig (Other); University Hospital, Antwerp (Other); Medical University of Graz (Other); Norwegian University of Science and Technology (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EU 602405-2
Record Dates: First submitted 2014-02-25; First posted 2014-03-05 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Diastolic heart failure, Heart failure with preserved ejection fraction, exercise
MeSH Terms: conditions — Heart Failure, Diastolic; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Intensity Exercise (Experimental): Patients perform interval- type endurance exercise at high intensity
  Interventions: Behavioral: High Intensity Exercise
- Moderate Continuous Exercise (Active Comparator): Patients perform endurance exercise at moderate intensity
  Interventions: Behavioral: Moderate Continuous Exercise
- Usual Care (Sham Comparator): Patients receive advice on being physically active as well as usual care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: High Intensity Exercise
  Arms: High Intensity Exercise
Behavioral: Moderate Continuous Exercise
  Arms: Moderate Continuous Exercise
Behavioral: Usual Care
  Arms: Usual Care

SUMMARY:
Aim of the clinical multicenter study (OptimEx-CLIN) is to assess the optimal exercise intervention in patients with Heart Failure with preserved Ejection Fraction (HFpEF; also termed diastolic heart failure) that will best improve peak oxygen uptake (Peak Vo2) and additionally diastolic function (assessed echocardiographically). The investigators hypothesize that exercise training reverses HFpEF and that intensity of exercise training is more important than duration.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (structured exercise < 2x 30 min/wk)
* At least 40 years old
* Preserved systolic function LVEF > 50%
* Signs and symptoms of heart failure class NYHA II or III
* Diastolic dysfunction (E/é > 15 or E/é 8-15 and NT-proBNP > 220 pg/ml)
* Clinically stable for >= 6 weeks
* Optimal medical treatment for >= 6 weeks
* Written informed consent

Exclusion Criteria:

* Non- HFpEF causes for HF symptoms (significant valvular or coronary disease, uncontrolled hypertension or arrhythmias, primary cardiomyopathies)
* Significant pulmonary disease (FEV1 < 50% predicted, COPD GOLD III-IV)
* Inability to exercise or conditions that may interfere with exercise intervention
* Myocardial infarction in the previous three months
* Signs of ischemia during exercise testing
* Comorbidity that may influence one- year prognosis
* Participation in another clinical trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Change in Peak VO2 after three months | Baseline and three months
  Change in Peak VO2 after three month intervention

SECONDARY OUTCOMES:
Change in E/e' (representing diastolic filling pressure) at baseline and three months | three months
  Change in E/e' (representing diastolic filling pressure) at baseline and three months
Change in E/e' at baseline and 12 months | 12 months
  Change in E/e' at baseline and 12 months
Change in Peak VO2 at baseline and 12 months | 12 months
  Change in Peak VO2 at baseline and 12 months
Change in NTproBNP at baseline and three months | three months
  Change in NTproBNP at baseline and three months
Change in NTproBNP at baseline and 12 months | 12 months
  Change in NTproBNP at baseline and 12 months
Change in health related quality of life at baseline and three months | three months
  Change in HRQOL as measured by the Kansas City Cardiomyopathy Questionnaire at baseline and three months
Change in health related Quality of life at baseline and 12 months | 12 months
  Change in HRQOL as measured by the Kansas City Cardiomyopathy Questionnaire at baseline and 12 months
Change in Left Atrial Volume Index (LAVI) at baseline and three months | three months
  Change in Left Atrial Volume Index (LAVI) at baseline and three months
Change in Left Atrial Volume Index (LAVI) at baseline and 12 months | 12 months
  Change in Left Atrial Volume Index (LAVI) at baseline and 12 months
Change in e' medial at baseline and three months | three months
  Change in e' medial at baseline and three months
Change in e' at baseline and 12 months | 12 months
  Change in e' at baseline and 12 months
Change in submaximal exercise capacity at baseline and three months | three months
  submaximal exercise capacity will be measured using watts at the first ventilatory threshold (VT1)
Change in submaximal exercise capacity at baseline and 12 months | 12 months
  Submaximal exercise capacity will be measured using watts at the first ventilatory threshold (VT1)
Change in VE/VCO2 slope at baseline and three months | three months
  Change in VE/VCO2 slope at baseline and three months
Change in VE/VCO2 slope at baseline and 12 months | 12 months
  Change in VE/VCO2 slope at baseline and 12 months
Change in Flow Mediated Dilation (FMD) at baseline and three months | three months
  Change in Flow Mediated Dilation (FMD) at baseline and three months
Change in Flow Mediated Dilation (FMD) at baseline and 12 months | 12 months
  Change in Flow Mediated Dilation (FMD) at baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, M.D., Study Director — Technische Universität München, Munich, Germany; Martin Halle, M.D., Principal Investigator — Technische Universität München, Munich, Germany; Burkert Pieske, M.D., Principal Investigator — Charite University, Berlin, Germany; Christiaan Vrints, M.D., Principal Investigator — Antwerp University Hospital, Belgium; Volker Adams, Ph.D., Principal Investigator — Heart Center Leipzig, Leipzig, Germany; Ulrik Wisløff, Ph.D., Principal Investigator — Norwegian University of Science and Technology, Trondheim, Norway; Axel Linke, M.D., Principal Investigator — Heart Center Leipzig, Leipzig, Germany; Frank Edelmann, M.D., Principal Investigator — Charite University, Berlin, Germany
Locations (4):
- Department of Cardiology, Antwerp University Hospital, Edegem, Belgium
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinik für Innere Medizin/ Kardiologie, Herzzentrum Leipzig- Universitätsklinik, Leipzig
  - Department of Prevention, Rehabilitation and Sports Medicine, Technische Universität München, Munich

REFERENCES:
- [Result] Gevaert AB, Witvrouwen I, Van Craenenbroeck AH, Van Laere SJ, Boen JRA, Van de Heyning CM, Belyavskiy E, Mueller S, Winzer E, Duvinage A, Edelmann F, Beckers PJ, Heidbuchel H, Wisloff U, Pieske B, Adams V, Halle M, Van Craenenbroeck EM; OptimEx-Clin Study Group. miR-181c level predicts response to exercise training in patients with heart failure and preserved ejection fraction: an analysis of the OptimEx-Clin trial. Eur J Prev Cardiol. 2021 Dec 29;28(15):1722-1733. doi: 10.1093/eurjpc/zwab151. PMID 34508569
- [Result] Mueller S, Haller B, Halle M; OptimEx-Clin Study Group. Effect of Training on Peak Oxygen Consumption in Patients With Heart Failure With Preserved Ejection Fraction-Reply. JAMA. 2021 Aug 24;326(8):772-773. doi: 10.1001/jama.2021.10061. No abstract available. PMID 34427605
- [Derived] Gevaert AB, Bohm B, Hartmann H, Goovaerts I, Stoop T, Van De Heyning CM, Beckers PJ, Baldassarri F, Mueller S, Oberhoffer R, Duvinage A, Haykowsky MJ, Wisloff U, Adams V, Pieske B, Halle M, Van Craenenbroeck EM. Effect of Training on Vascular Function and Repair in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2023 Apr;11(4):454-464. doi: 10.1016/j.jchf.2022.12.011. Epub 2023 Mar 1. PMID 36892488
- [Derived] Winzer EB, Augstein A, Schauer A, Mueller S, Fischer-Schaepmann T, Goto K, Hommel J, van Craenenbroeck EM, Wisloff U, Pieske B, Halle M, Linke A, Adams V. Impact of Different Training Modalities on Molecular Alterations in Skeletal Muscle of Patients With Heart Failure With Preserved Ejection Fraction: A Substudy of the OptimEx Trial. Circ Heart Fail. 2022 Oct;15(10):e009124. doi: 10.1161/CIRCHEARTFAILURE.121.009124. Epub 2022 Oct 6. PMID 36200450
- [Derived] Gevaert AB, Mueller S, Winzer EB, Duvinage A, Van de Heyning CM, Pieske-Kraigher E, Beckers PJ, Edelmann F, Wisloff U, Pieske B, Adams V, Halle M, Van Craenenbroeck EM; OptimEx-Clin Study Group. Iron Deficiency Impacts Diastolic Function, Aerobic Exercise Capacity, and Patient Phenotyping in Heart Failure With Preserved Ejection Fraction: A Subanalysis of the OptimEx-Clin Study. Front Physiol. 2022 Feb 10;12:757268. doi: 10.3389/fphys.2021.757268. eCollection 2021. PMID 35222057
- [Derived] Mueller S, Winzer EB, Duvinage A, Gevaert AB, Edelmann F, Haller B, Pieske-Kraigher E, Beckers P, Bobenko A, Hommel J, Van de Heyning CM, Esefeld K, von Korn P, Christle JW, Haykowsky MJ, Linke A, Wisloff U, Adams V, Pieske B, van Craenenbroeck EM, Halle M; OptimEx-Clin Study Group. Effect of High-Intensity Interval Training, Moderate Continuous Training, or Guideline-Based Physical Activity Advice on Peak Oxygen Consumption in Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2021 Feb 9;325(6):542-551. doi: 10.1001/jama.2020.26812. PMID 33560320
- [Derived] Suchy C, Massen L, Rognmo O, Van Craenenbroeck EM, Beckers P, Kraigher-Krainer E, Linke A, Adams V, Wisloff U, Pieske B, Halle M. Optimising exercise training in prevention and treatment of diastolic heart failure (OptimEx-CLIN): rationale and design of a prospective, randomised, controlled trial. Eur J Prev Cardiol. 2014 Nov;21(2 Suppl):18-25. doi: 10.1177/2047487314552764. PMID 25354950
- See also: Related Info — http://www.ntnu.edu/optimex